CLINICAL TRIAL: NCT03561298
Title: An Open-label, Fixed-Sequence Study in Healthy Male Subjects to Assess the Drug Interaction Potential of Multiple Doses of Zanubrutinib With a Drug "Cocktail" Representative for CYP3A4, CYP2C9, CYP2C19, P-gP and BCRP Substrates
Brief Title: A Pharmacokinetic Study to Assess Drug-drug Interaction Between Zanubrutinib and a Cocktail of Substrates in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-108
Record Dates: First submitted 2018-05-24; First posted 2018-06-19 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2018-10

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; Healthy subjects
MeSH Terms: interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm: BGB-3111 + Drug Cocktail (Experimental): BGB-3111 and Drug Cocktail (midazolam, warfarin, omeprazole, digoxin and rosuvastatin)
  Interventions: Drug: BGB-3111 and Drug Cocktail

INTERVENTIONS:
Drug: BGB-3111 and Drug Cocktail — BGB-3111 and Drug Cocktail (midazolam, warfarin, omeprazole, digoxin and rosuvastatin)

SUMMARY:
This study is designed to evaluate the safety and pharmacokinetic interaction of effects of multiple doses of zanubrutinib with a "Cocktail" of five probe drugs for cytochrome P450 (CYP) 3A, CYP2C9, CYP2C19, P-glycoprotein and breast cancer resistance protein (BCRP) in healthy subjects

ELIGIBILITY:
Inclusion Criteria: All Groups

* Male subjects in good health as determined by past medical history, physical examination, vital signs, ECG and laboratory tests at screening.
* Subjects must have a body mass index (BMI) between 18 and 32 kg/m2.
* Male subjects must agree to a highly effective method of birth control from screening until at least 90 days after the last dose of study drug.

Exclusion Criteria:

* Subjects with a clinically relevant history or presence of any clinically significant disease.
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy, cholecystectomy, and hernia repair will be allowed).
* History of drug or alcohol abuse within 2 years prior to Check-In.
* Alcohol consumption of >21 units per week.
* A positive urine drug screen and/or positive alcohol breath test at Screening and/or Check-in.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result and/or a positive human immunodeficiency virus (HIV) at screening.
* Use of tobacco- or nicotine-containing products within 3 months prior to Check-In.
* History of blood donation of 56 days prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
PK parameters of probe drugs (warfarin, midazolam, digoxin, rosuvastatin, and omeprazole) derived from the plasma concentration time profile before and after oral administration of zanubrutinib | Days 1-20
  AUC from time 0 to the last quantifiable concentration (AUC0-t)
PK parameters of probe drugs (warfarin, midazolam, digoxin, rosuvastatin, and omeprazole) derived from the plasma concentration time profile before and after oral administration of zanubrutinib | Days 1-20
  AUC from time 0 to infinity (AUC0 ∞; calculated as appropriate and allowed by the available data)
PK parameters of probe drugs (warfarin, midazolam, digoxin, rosuvastatin, and omeprazole) derived from the plasma concentration time profile before and after oral administration of zanubrutinib | Days 1-20
  Maximum observed plasma concentration (Cmax)
PK parameters of probe drugs (warfarin, midazolam, digoxin, rosuvastatin, and omeprazole) derived from the plasma concentration time profile before and after oral administration of zanubrutinib | Days 1-20
  Time of the maximum observed plasma concentration (Tmax)

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability. | up to 26 days
  An adverse event is an unfavorable and unintended sign (including an abnormal laboratory finding, an abnormal electrocardiogram), symptom or disease (new or exacerbated) temporally associated with the use of a study drug, whether considered related to study drug or not.

CONTACTS AND LOCATIONS:
Overall Officials: William Novotny, MD, Study Director — BeiGene
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No